CLINICAL TRIAL: NCT02919072
Title: Comparison of Epidural Chloroprocaine 3% and Ropivacaine 0.75% for Unplanned Caesarean Section in Labouring Women Who Have an Epidural Catheter in Situ
Brief Title: Chloroprocaine 3% - Epidural Anesthesia in Unplanned Caesarean Section
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The doctors involved in the study did not enroll any patients
Sponsor: Sintetica SA (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHL.3/01-2016
Record Dates: First submitted 2016-08-29; First posted 2016-09-29 (Estimated); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Unplanned Caesarean Section
MeSH Terms: interventions — chloroprocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroprocaine (Experimental): Chloroprocaine, 20 ml epidural anaesthetic solution administered according to the standard procedures of the hospital. In case of pain or discomfort, a 6 mL epidural top-up will be administered.
  Interventions: Drug: Chloroprocaine
- Ropivacaine (Active Comparator): Ropivacaine, 20 ml epidural anaesthetic solution administered according to the standard procedures of the hospital. In case of pain or discomfort, a 6 mL epidural top-up will be administered.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Chloroprocaine — The 20 mL epidural anaesthetic solution will be administered as follows: 5 mL of the study anaesthetic solution will be given epidurally and the block will be assessed after 2 minutes from the first injection using cold, pinprick and touch. Then intrathecal placement will be excluded and a further 15 mL of the study anaesthetic solution will be administered epidurally. Two minutes after the start of the second injection, the sensory block will be re-assessed using cold, pinprick and touch. In case of pain or discomfort a 6 mL epidural top-up of the same anaesthetic will be administered.
  Other Names: Ampres
  Arms: Chloroprocaine
Drug: Ropivacaine — The 20 mL epidural anaesthetic solution will be administered as follows: 5 mL of the study anaesthetic solution will be given epidurally and the block will be assessed after 2 minutes from the first injection using cold, pinprick and touch. Then intrathecal placement will be excluded and a further 15 mL of the study anaesthetic solution will be administered epidurally. Two minutes after the start of the second injection, the sensory block will be re-assessed using cold, pinprick and touch. In case of pain or discomfort a 6 mL epidural top-up of the same anaesthetic will be administered.
  Other Names: Naropin
  Arms: Ropivacaine

SUMMARY:
The study evaluate the quality of epidural anaesthesia and the safety of Chloroprocaine HCl 3% compared with Ropivacaine HCl 0.75% in patients with an epidural catheter in situ undergoing unplanned Caesarean section.

DETAILED DESCRIPTION:
Labouring women who have an epidural catheter in situ and established analgesia, in need of an unplanned Caesarean section, will be randomly allocated to receive either Chloroprocaine HCl 3% (T-group) or Ropivacaine HCl 0.75% (R-group) epidurally. Prior to the epidural injection, the patient will be transferred to the operating theatre. The local anaesthetic solution will be freshly prepared and 20 mL will be administered by epidural injection, according to the standard hospital procedures, as detailed in the "Study Schedule" section below. Time T0 is defined as the start time of the first epidural injection of the investigational product. In case of pain or discomfort, a 6 mL epidural top-up of the same anaesthetic, i.e. Chloroprocaine HCl 3% in T-group and Ropivacaine HCl 0.75% in R-group, will be administered. The anaesthesiologist(s) administering the anaesthetic and collecting the data will be blinded with respect to the treatment given to each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: Signed written informed consent before inclusion in the study (obtained from women fulfilling the criteria, only when effective analgesia has been established)
2. Sex, pregnancy status and age: Labouring women with singleton pregnancy, ≥ 18 years old
3. Epidural catheter: Previously sited epidural catheter
4. ASA physical status: I-II
5. Analgesia: Effective analgesia established following combined spinal epidural analgesia (CSE)
6. Term gestation: ≥ 36 weeks
7. Caesarean section: Unplanned Caesarean section category 2 or 3, according to Lucas Classification
8. Body Mass Index (BMI): ≤ 40 kg/m2
9. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Physical findings: Clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to epidural anaesthesia
2. ASA physical status: III-V
3. Further anaesthesia: Patients expected to require further anaesthesia
4. Epidural catheter: Epidural catheter failure (epidural catheter replacement required or inability to provide effective analgesia)
5. Pregnancy: Labouring women with multiple pregnancy
6. Caesarean section: Elective Caesarean section
7. Allergy: ascertained or presumptive hypersensitivity to the active principle and /or formulations ingredients; ascertained or presumptive hypersensitivity to the amide and ester-type anaesthetics
8. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric diseases, eclampsia, antepartum haemorrhage, sepsis, blood coagulation disorders, insulin dependent diabetes mellitus, terminal kidney failure
9. Medications: Medication known to interfere with the extent of regional blocks (see chloroprocaine and ropivacaine SmPCs) for 2 weeks before the start of the study
10. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study
11. Drug, alcohol: history of drug or alcohol abuse
12. Plasma cholinesterase: Known plasma cholinesterase deficiency.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Van de Velde, MD, Principal Investigator — Department of Anesthesiology, UZ Leuven, campus Gasthuisberg
Locations (1):
- UZ Leuven, campus Gasthuisberg, Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to difficulties in enrolling patients, the enrolment stopped prematurely, and only 16 patients were screened and randomised (only at site N. 001).
Period: Overall Study
Arm/Group | Chloroprocaine | Ropivacaine
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroprocaine | Ropivacaine | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (5.6) | 33.3 (7.5) | 31.05 (6.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Time to the Onset of Anaesthesia
Description: The time from T0 (start time of the epidural injection) to complete loss of cold sensation to the metameric level T4 (block to T4), bilateral.
Time Frame: Up to 1 hour after last epidural injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Ropivacaine
Number analyzed (Participants) | 6 | 7
minutes | 9 (5.8) | 9.1 (4)

2. Secondary Outcome: Time From T0 to Loss Light Touch Sensation
Description: Time from T0 to loss light touch sensation to the metameric level T5 (block to T5), bilateral
Time Frame: Up to 1 hour after last epidural injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Chloroprocaine | Ropivacaine
Number analyzed (Participants) | 3 | 6
minutes | 9.3 (9.2) | 13.3 (4.1)

3. Secondary Outcome: Quality of the Block
Description: Quality of the block assessed between 10 and 20 min after the end of surgery by the anaesthesiologist and patient together using a 0-10 cm visual analogue scale (VAS; 10=excellent anaesthetic quality, 0=very poor anaesthetic quality)
Time Frame: Quality of the block assessed between 10 and 20 minutes after the end of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chloroprocaine | Ropivacaine
Number analyzed (Participants) | 6 | 7
units on a scale | 9.8 (0.4) | 8.4 (3.7)

4. Secondary Outcome: Maximum Metameric Level of the Sensory Block
Description: Maximum metameric level of the sensory block assessed by three modalities (complete loss of cold, pinprick and light touch sensation)
Time Frame: Up to 1 hrs after last epidural injection
Reporting Status: Not Posted

5. Secondary Outcome: Motor Block Assessment
Description: Motor block assessment (modified Bromage scale) at baseline, prior to incision and after surgery
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Patients Who Need Top-up Anaesthesia
Description: Proportion of patients who need top-up epidural anaesthesia (same anaesthetic as first epidural injection)
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Patients Who Need Supplementation of Opioids
Description: Proportion of patients who need supplementation of the block intraoperatively with intravenous opioids
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

8. Secondary Outcome: Proportion of Patients Who Need General Anaesthesia
Description: Proportion of patients who need general anaesthesia
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

9. Secondary Outcome: Discomfort and Pain During Surgery
Description: Discomfort and pain assessed during surgery through spontaneous patient's reporting and questioning by the Investigator/anaesthesiologist
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

10. Secondary Outcome: First Breakthrough Pain
Description: First breakthrough pain assessed by the patient, recorded on a 0-10 cm VAS (0=no pain, 10= most severe pain imaginable)
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

11. Secondary Outcome: Maternal Treatment-emergent Adverse Events
Description: Maternal treatment-emergent adverse events, with particular attention to pain (see above), pruritus, nausea, vomiting
Time Frame: Up to day 3±1 after surgery
Reporting Status: Not Posted

12. Secondary Outcome: Pulse Rate
Description: Maternal pulse rate
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

13. Secondary Outcome: Oximetry
Description: Maternal pulse oximetry (SpO2)
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

14. Secondary Outcome: Electrocardiogram
Description: Maternal electrocardiogram
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

15. Secondary Outcome: Total Dose of Phenylephrine
Description: Total dose (μg) of phenylephrine
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

16. Secondary Outcome: Total Dose of Atropine
Description: Total dose (mg) of atropine
Time Frame: Up to 2 hours after last epidural injection
Reporting Status: Not Posted

17. Secondary Outcome: Intravenous Fluids
Description: Total volume (ml) of intravenous fluids
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

18. Secondary Outcome: Neonate Apgar
Description: Neonate Apgar scores at 1 and 5 minutes
Time Frame: 1 and 5 minutes after birth
Reporting Status: Not Posted

19. Secondary Outcome: Foetal Hypoxic Stress
Description: Indication of foetal hypoxic stress
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

20. Secondary Outcome: Pain at the Site of Surgery
Description: Pain at the site of surgery at final visit/early termination visit, recorded on a 0-10 cm VAS (0=no pain, 10=most severe pain imaginable)
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

21. Secondary Outcome: Pain at the Site of Epidural Injection
Description: Pain at the site of epidural injection at final visit/early termination visit, recorded on a 0-10 cm VAS (0=no pain, 10=severe pain)
Time Frame: Up to 12 hours after surgery
Reporting Status: Not Posted

22. Secondary Outcome: Concomitant Medications
Description: Maternal concomitant medications
Time Frame: Up to day 3±1 after surgery
Reporting Status: Not Posted

23. Secondary Outcome: Neonatal Adverse Events
Description: Neonatal adverse events
Time Frame: Up to day 3±1 after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Maternal AEs will be assessed throughout the study from the signature of the informed consent up to follow-up Visit Day 3±1
Arm/Group | Chloroprocaine | Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chloroprocaine (N=8) | Ropivacaine (N=8)
Hypotensio (Vascular disorders) | 5 (5) | 7 (8)
post lumbar puncture syndrom (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POst procedural disconfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT02919072/Prot_SAP_000.pdf